CLINICAL TRIAL: NCT03529760
Title: Chemotherapy Efficacy and Follow-up Study of Hepatitis B Virus Infection and Reactivation in Children With Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qiu Li, Director, Children's Hospital of Chongqing Medical University
Other Study IDs: 2018-27
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Reactivation of Hepatitis B Virus
Keywords: Leukemia, occult hepatitis B virus infection
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Separating serum, stored at -80 degrees Celsius
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children with clinically diagnosed leukemia may experience occult HBV infection after chemotherapy immunosuppressive therapy, which may affect the normal course of leukemia treatment. However, this is not caused by clinically relevant diagnosis and treatment measures but exists in vivo.

DETAILED DESCRIPTION:
The clinical diagnosis of children with leukemia may be due to the influence of leukemia disease on the immune cells of the children and the damage to the immune system due to immunosuppressive therapy in children. Therefore, the risk of contracting hepatitis B virus is relatively high, and some children are In the treatment of immunosuppressive chemotherapy (later), the reactivation of occult HBV infection has an impact on the normal course of leukemia treatment. However, this is not a clinically relevant diagnosis and treatment measure. It is necessary to avoid unnecessary conflicts between clinical doctors and patients as much as possible.

ELIGIBILITY:
Inclusion Criteria:

The clinical diagnosis of children with leukemia received systemic chemotherapy.

Exclusion Criteria:

Children with non-leukemia and children without appropriate treatment.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1-16-year-old leukemia hospitalized chemotherapy children
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-07-15 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
HBV-DNA positive | 1-year
  Positive HBV nucleic acid test

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, Study Director — Chongqing Children's Hospital of Chongqing Medical University
Locations (1):
- Chongqing Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China